CLINICAL TRIAL: NCT02386020
Title: Clinical Efficacy of Locally Delivered Aloe Vera Gel as an Adjunct to Non-surgical Periodontal Therapy in Chronic Periodontitis Subjects With Type 2 Diabetes Mellitus: a Randomized Controlled Clinical Trial
Brief Title: Aloe Vera in Chronic Periodontitis With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Government Dental College and Research Institute, Bangalore (Other)
Responsible Party: Principal Investigator, Dr. A R Pradeep, Professor & Head, Department of Periodontology, Government Dental College and Research Institute, Bangalore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GDCRI/ACM/PG/PhD/10E/2013-14
Record Dates: First submitted 2015-02-18; First posted 2015-03-11 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-02

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): After SRP, placebo gel was delivered subgingivally into periodontal pockets.
  Interventions: Drug: placebo gel
- Aloe vera (Active Comparator): After SRP, aloe vera gel was delivered subgingivally into periodontal pockets.
  Interventions: Drug: aloe vera

INTERVENTIONS:
Drug: aloe vera — After SRP, aloe vera gel was delivered subgingivally into periodontal pockets.
  Arms: Aloe vera
Drug: placebo gel — After SRP, placebo gel was delivered subgingivally into periodontal pockets.
  Arms: Placebo

SUMMARY:
The present study is designed to investigate the effectiveness of AV gel local drug delivery as an adjunct to scaling and root planing (SRP) in the treatment of subjects with chronic periodontitis (CP) and type 2 diabetes mellitus (DM).

DETAILED DESCRIPTION:
BACKGROUND: Advances in the field of alternative medicine have promoted widespread use of herbal agents, like Aloe vera (AV), for both medical and dental therapy. AV has anti-inflammatory, antioxidant, antimicrobial, hypoglycaemic, healing promoting and immune boosting properties. The present study is designed to investigate the effectiveness of AV gel local drug delivery as an adjunct to scaling and root planing (SRP) in the treatment of subjects with chronic periodontitis (CP) and type 2 diabetes mellitus (DM).

MATERIAL AND METHODS: A total of 60 subjects with probing depth (PD) ≥5mm and clinical attachment level (CAL) ≥3mm were randomly divided into two groups. Group 1 was treated with SRP + placebo gel local drug delivery (LDD) and Group 2 with SRP + AV gel LDD. Clinical parameters including full mouth plaque index (PI), modiﬁed sulcus bleeding index (mSBI), probing depth (PD) and clinical attachment level (CAL) were recorded first at baseline and then at intervals of 3 months and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Well-controlled type 2 DM
* Chronic periodontitis with moderate to deep pockets [probing depth (PD) ≥5mm and clinical attachment loss (CAL) ≥3mm]
* No history of antibiotic or periodontal therapy in the preceding 6 months.

Exclusion Criteria:

* Any known disease/condition or on any medication that can affect the periodontal status
* Known or suspected allergy to herbal medications
* Systemic antimicrobial therapy
* Aggressive periodontitis
* Smokers
* Alcoholics
* Immunocompromised patients
* Pregnant or lactating females

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in Clinical attachment level | baseline to 6 months

SECONDARY OUTCOMES:
Change in Plaque index | baseline to 6 months
Change in modified sulcus bleeding index | baseline to 6 months
Change in Probing depth | baseline to 6 months